CLINICAL TRIAL: NCT00714584
Title: Pharmacokinetics of Naltrexone Hydrochloride (HCl) Following Intravenous (i.v.) and Oral Routes of Administration in Healthy Subjects
Brief Title: Pharmacokinetics of Naltrexone Following Intravenous and Oral Routes of Administration in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alza Corporation, DE, USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR003256
Record Dates: First submitted 2008-07-10; First posted 2008-07-14 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-04

CONDITIONS: Biological Availability
Keywords: Infusions, Intravenous; Safety; Pharmacokinetics; Naltrexone; Administration, Oral
MeSH Terms: interventions — Naltrexone

INTERVENTIONS:
Drug: Naltrexone HCl.

SUMMARY:
The purpose of the study is to compare the pharmacokinetics of naltrexone following i.v. and oral administration in healthy volunteers, and to assess the bioavailability of naltrexone following oral administration. Moreover, safety is assessed.

DETAILED DESCRIPTION:
Naltrexone blocks the effects of opioid (morphine-like) drugs by competitive binding at the opioid receptors in the brain. Naltrexone does not possess morphine-like properties and exhibits minimal pharmacologic activity. Naltrexone is marketed as an oral tablet. A wide range of oral bioavailability values have been reported for naltrexone. The wide range in oral bioavailability of naltrexone appears to be due to differences in assay specificity and the method of estimation of bioavailability (use of total drug, free drug, or urinary excretion data rather than plasma level). This was a single-center, randomized (study drug assigned by chance), open-label, 2-treatment, 2-period crossover study in healthy volunteers. Healthy volunteers were randomly assigned to 1 of 2 treatment sequences (AB or BA) with a washout period of 6 to 14 days between treatments. The washout period commenced the day of dosing, after drug administration. Blood samples for determination of blood naltrexone levels were collected at scheduled time points from the arm opposite to the 1 selected for naltrexone i.v. administration. Pulse, blood pressure, breathing rate, body temperature were measured at the times listed in the study schema. Healthy volunteers remained at the research facility for blood sample collection periods and were monitored for adverse events throughout the treatment periods.

Treatment A: 1 mg naltrexone HCl administered i.v. over 15 minutes (naltrexone i.v.). Treatment B: 50 mg naltrexone HCl administered orally (naltrexone oral).

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non smoker, men and nonpregnant nonlactating women
* Weighing a minimum of 60 kg and were within 15% of ideal weight for height as described in the Metropolitan Life Insurance Height and Weight Standards
* Who did not have a history or show presence of drug or alcohol dependence or abuse

Exclusion Criteria:

* Known allergy or hypersensitivity to naltrexone
* Usage of prescription medication including opioids (except for birth control medications, sex-hormone replacement, vitamins) within 14 days prior to Day 1, over-the-counter medication (except for vitamin supplements or acetaminophen [less than 2 g/day]) or herbal medication within 3 days prior to Day 1, alcohol, grapefruit juice, or caffeine within 48 hours before dosing
* Consumption of more than 450 mg of caffeine per day (eg, approximately 5 cups of tea, 3 cups of regular coffee, or 8 cans of cola)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2003-05; Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Evaluate the pharmacokinetics of naltrexone following i.v. and oral routes of administration in healthy volunteers, and to assess the absolute bioavailability of naltrexone following oral administration.

SECONDARY OUTCOMES:
Assessment of safety. Vital signs, Physical examination, clinical laboratory tests, and electrocardiogram were performed at screening and study termination. Additionally, vital signs were recorded on Days 1 and 2 of both treatment periods.

CONTACTS AND LOCATIONS:
Overall Officials: Alza Corporation Clinical Trial, Study Director — Alza Corporation, DE, USA

REFERENCES:
- See also: Pharmacokinetics of naltrexone following intravenous and oral routes of administration in healthy subjects — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=91&filename=CR003256_CSR.pdf